CLINICAL TRIAL: NCT06731790
Title: Role of the Nuclear Pore Component RANBP2 in Inflammatory Responses to Viral Infections
Acronym: InflammaNUP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Institut de Recherche en Infectiologie de Montpellier (CNRS) (Unknown); A*STAR Infectious Diseases Labs (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RECHMPL23_0455
Record Dates: First submitted 2024-12-09; First posted 2024-12-12 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-11

CONDITIONS: Rare Genetic Disease; Acute Necrotizing Encephalopathy
Keywords: RANBP2; nuclear pore
MeSH Terms: conditions — Leukoencephalitis, Acute Hemorrhagic | interventions — Blood Specimen Collection; Genetic Testing

STUDY DESIGN:
Intervention Model Description: Controlled, pathophysiological, exploratory interventional pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mutant RANBP2 associated with predisposition to ANE1 (Experimental): Subjects aged 1 to 90 with a T585M mutation in RANBP2 for the "RANBP2 mutation" arm. During a single visit, 2 tubes of blood will be sampled, demographic data and clinical history collected, and a clinical examination performed.
  Interventions: Other: Blood sampling for inflammatory phenotype analysis; Genetic: Blood sampling for genetic analysis
- Healthy control subjects (Active Comparator): For healthy control subjects related to a person from the "mutant RANBP2" arm: During a single visit, 2 tubes of blood will be sampled, demographic data and clinical history collected, and a clinical examination performed. Healthy control subjects related to a person from the "mutant RANBP2" arm will be included in the third Secondary Outcome (whole exome sequencing).
  For healthy control subjects unrelated to a person from the "mutant RANBP2" arm: During a routine epilepsy consultation for children, or a family disease screening for adults, an additional blood tube will be sampled, demographic data collected and a clinical examination performed. Healthy control subjects unrelated to a person from the "mutant RANBP2" arm will not be included in the third Secondary Outcome (whole exome sequencing).
  Interventions: Other: Blood sampling for inflammatory phenotype analysis; Genetic: Blood sampling for genetic analysis

INTERVENTIONS:
Other: Blood sampling for inflammatory phenotype analysis — Blood sampling for basal and post-stimulation inflammatory phenotype analysis
Genetic: Blood sampling for genetic analysis — Collection of a blood tube for whole exome sequencing, , long-read sequencing of the RANBP2 gene and analysis of the presence of the mutation by RTqPCR.

SUMMARY:
The goal of this controlled, pathophysiological, exploratory interventional study is to compare the inflammatory phenotype of circulating immune cells, basal and following stimulation, from Acute Necrotizing Encephalopathy Type 1 (ANE1) patients with those from sex- and age-matched donors who do not carry the mutation.To date, no study has investigated the molecular mechanisms regulating the inflammatory response in ANE1 disease directly on patient samples.

The primary endpoint in individuals in the "mutated RANBP2" arm is an inflammatory phenotype (hyperinflammatory monocytes, secretion of pro-inflammatory cytokines, anti-glycoprotein autoantibodies), significantly exacerbated basal and/or post-stimulation production of pro-inflammatory cytokines compared with the control arm.

The secondary objective is to examine the allelic expression of mutant RANBP2 and characterize genetic variants by whole-exome sequencing, in order to associate them with RANBP2 protein localization and ANE crisis severity

The researchers will compare the group of ANE1 patients with age- and sex-matched control groups, divided into two subgroups: unrelated controls and controls with familial ties. The aim is to study the different types of inflammatory responses and correlate them with the localization of the RANBP2 protein and the severity of ANE episodes.

Participants will participate in a single visit during which demographic data, clinical history and a blood test will be collected with one (unrelated control) or two blood tubes (ANE1 and related control).

DETAILED DESCRIPTION:
The nucleoporin RANBP2, also known as Nup358, is a component of the cytoplasmic filaments of nuclear pore complexes (NPCs), which regulate the transport of macromolecules between the cytoplasm and the nucleus. Mutations in the RANBP2 gene are associated with a rare genetic predisposition to acute necrotizing encephalopathy (ANE1), a predominantly pediatric disease characterized by multiple, symmetrical hemorrhagic lesions of the brain following febrile infection, most often with influenza A virus (IAV). Given the presumed inflammatory nature of ANE1, first-line treatment includes intravenous administration of high-dose pharmacological corticosteroids with or without immunoglobulins. In addition, two clinical cases report that IL-6 inhibition by tocilumizab may have a beneficial role.

The research team have recently demonstrated that loss or mislocalisation of RANBP2, as seen with ANE-linked mutations, boosts influenza virus replication and triggers excessive inflammation.

The researchers hypothesis is that mutation of RANBP2 in ANE1 patients weakens nuclear pore control of innate immune signaling pathways, leading to an exacerbated inflammatory response to infections.

ELIGIBILITY:
Inclusion Criteria:

* Obtaining written consent from adult participants
* Obtaining written consent from legal guardians of minors with their assent
* Subjects aged 1 to 90
* Subject with a T585M mutation in RANBP2 for the RANBP2 mutation arm.
* Subjects matched on age (+/- 10 years) and gender for the "control" arm.

Exclusion Criteria:

* Patient not affiliated to a social security scheme or not a beneficiary of such a scheme. (for example, a European Health Insurance Card (EHIC))
* Absence of written informed consent
* Person unable to give consent
* legally protected adult (guardianship, curatorship)
* Person deprived of liberty
* Person participating in another research study with an exclusion period still in progress

Ages: 1 Year to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2025-04-24 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Comparison of the inflammatory phenotype of circulating immune cells, both basal and following stimulation, from ANE1 patients with those from sex- and age-matched donors not carrying the mutation | Baseline
  These experiments will be carried out on blood, serum, peripheral blood mononuclear cells (PBMC) and monocyte-derived macrophages and microglia (MDM and MMG, respectively).
  The primary endpoint for individuals in the "mutated RANBP2" arm is an inflammatory phenotype, basal and/or after stimulation, that is significantly exacerbated compared with the "control" arms. Samples will be analyzed by ELISA/Luminex and flow cytometry. The expected difference will be a 2 to 10-fold upregulation in one or several markers of hyperinflammatory monocytes, and/or in one or several secreted pro-inflammatory cytokines, and/or in one or several autoantibodies, based on our results in PBMC treated with RANBP2-targeted RNA interference

SECONDARY OUTCOMES:
Determination of the allelic expression of mutated RANBP2 | Baseline
  The first secondary endpoint will be heterozygous expression of mutated RANBP2 in individuals in the "mutated RANBP2" arm. The method of evaluation will be RT-PCR targeted to RANBP2, followed by quantitative PCR discriminating for the mutation, a diagnostic method recently introduced in the IRIM laboratory.
Determination of the effect of the T585M heterozygous mutation on RANBP2 localization | Baseline
  The second secondary outcome will be the significantly exacerbated basal and/or post-stimulation RANBP2 delocalization compared with the "control" arm. This will be tested on monocyte-derived macrophages by confocal microscopy.
Characterization of genetic variants that are significantly associated with ANE seizure severity | Baseline
  The third secondary endpoint will be the identification of genetic variants associated with the history of ANE episodes, if any, and their severity. The evaluation method will be whole exome sequencing, and long-read sequencing, only on participants from ANE families in the "control" and "mutated RANBP2" arms.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre MEYER, MD, Principal Investigator — Montpellier University Hospital
Locations (1):
- CHU Gui de Chauliac, Montpellier, Hérault, France

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Koh JC, Murugasu A, Krishnappa J, Thomas T. Favorable Outcomes With Early Interleukin 6 Receptor Blockade in Severe Acute Necrotizing Encephalopathy of Childhood. Pediatr Neurol. 2019 Sep;98:80-84. doi: 10.1016/j.pediatrneurol.2019.04.009. Epub 2019 Apr 25. PMID 31201070
- [Background] Bashiri FA, Al Johani S, Hamad MH, Kentab AY, Alwadei AH, Hundallah K, Hasan HH, Alshuaibi W, Jad L, Alrifai MT, Hudairi A, Al Sheikh R, Alenizi A, Alharthi NA, Abdelmagid TA, Ba-Armah D, Salih MA, Tabarki B. Acute Necrotizing Encephalopathy of Childhood: A Multicenter Experience in Saudi Arabia. Front Pediatr. 2020 Oct 9;8:526. doi: 10.3389/fped.2020.00526. eCollection 2020. PMID 33163461
- [Background] Okumura A, Mizuguchi M, Kidokoro H, Tanaka M, Abe S, Hosoya M, Aiba H, Maegaki Y, Yamamoto H, Tanabe T, Noda E, Imataka G, Kurahashi H. Outcome of acute necrotizing encephalopathy in relation to treatment with corticosteroids and gammaglobulin. Brain Dev. 2009 Mar;31(3):221-7. doi: 10.1016/j.braindev.2008.03.005. Epub 2008 May 5. PMID 18456443
- [Background] Mizuguchi M. Acute necrotizing encephalopathy of childhood: a novel form of acute encephalopathy prevalent in Japan and Taiwan. Brain Dev. 1997 Mar;19(2):81-92. doi: 10.1016/s0387-7604(96)00063-0. PMID 9105653
- [Background] Lim HY, Ho VP, Lim TC, Thomas T, Chan DW. Serial outcomes in acute necrotising encephalopathy of childhood: A medium and long term study. Brain Dev. 2016 Nov;38(10):928-936. doi: 10.1016/j.braindev.2016.05.002. Epub 2016 May 30. PMID 27256511
- [Background] Lee JH, Kim AJ, Kyong TY, Jang JH, Park J, Lee JH, Lee MJ, Kim JS, Suh YJ, Kwon SR, Kim CW. Evaluating the Outcome of Multi-Morbid Patients Cared for by Hospitalists: a Report of Integrated Medical Model in Korea. J Korean Med Sci. 2019 Jul 1;34(25):e179. doi: 10.3346/jkms.2019.34.e179. PMID 31243937
- [Background] Sell K, Storch K, Hahn G, Lee-Kirsch MA, Ramantani G, Jackson S, Neilson D, von der Hagen M, Hehr U, Smitka M. Variable clinical course in acute necrotizing encephalopathy and identification of a novel RANBP2 mutation. Brain Dev. 2016 Sep;38(8):777-80. doi: 10.1016/j.braindev.2016.02.007. Epub 2016 Feb 26. PMID 26923722
- [Background] Li J, Huo F, Wang S, Fan Y, Wu J, Zhang Z, Liu S, Wang Q. Recurrent infection triggered encephalopathy syndrome in a pediatric patient with RANBP2 mutation and severe acute respiratory syndrome coronavirus 2 infection. Pediatr Investig. 2023 Nov 19;7(4):290-296. doi: 10.1002/ped4.12406. eCollection 2023 Dec. PMID 38050538
- [Background] Jiang J, Wang YE, Palazzo AF, Shen Q. Roles of Nucleoporin RanBP2/Nup358 in Acute Necrotizing Encephalopathy Type 1 (ANE1) and Viral Infection. Int J Mol Sci. 2022 Mar 24;23(7):3548. doi: 10.3390/ijms23073548. PMID 35408907
- [Background] Levine JM, Ahsan N, Ho E, Santoro JD. Genetic Acute Necrotizing Encephalopathy Associated with RANBP2: Clinical and Therapeutic Implications in Pediatrics. Mult Scler Relat Disord. 2020 Aug;43:102194. doi: 10.1016/j.msard.2020.102194. Epub 2020 May 15. PMID 32426208
- [Background] Denier C, Balu L, Husson B, Nasser G, Burglen L, Rodriguez D, Labauge P, Chevret L. Familial acute necrotizing encephalopathy due to mutation in the RANBP2 gene. J Neurol Sci. 2014 Oct 15;345(1-2):236-8. doi: 10.1016/j.jns.2014.07.025. Epub 2014 Jul 18. PMID 25128471
- [Background] Neilson DE, Adams MD, Orr CM, Schelling DK, Eiben RM, Kerr DS, Anderson J, Bassuk AG, Bye AM, Childs AM, Clarke A, Crow YJ, Di Rocco M, Dohna-Schwake C, Dueckers G, Fasano AE, Gika AD, Gionnis D, Gorman MP, Grattan-Smith PJ, Hackenberg A, Kuster A, Lentschig MG, Lopez-Laso E, Marco EJ, Mastroyianni S, Perrier J, Schmitt-Mechelke T, Servidei S, Skardoutsou A, Uldall P, van der Knaap MS, Goglin KC, Tefft DL, Aubin C, de Jager P, Hafler D, Warman ML. Infection-triggered familial or recurrent cases of acute necrotizing encephalopathy caused by mutations in a component of the nuclear pore, RANBP2. Am J Hum Genet. 2009 Jan;84(1):44-51. doi: 10.1016/j.ajhg.2008.12.009. PMID 19118815
- [Background] Mizuguchi M, Abe J, Mikkaichi K, Noma S, Yoshida K, Yamanaka T, Kamoshita S. Acute necrotising encephalopathy of childhood: a new syndrome presenting with multifocal, symmetric brain lesions. J Neurol Neurosurg Psychiatry. 1995 May;58(5):555-61. doi: 10.1136/jnnp.58.5.555. PMID 7745402
- [Background] Desgraupes S, Etienne L, Arhel NJ. RANBP2 evolution and human disease. FEBS Lett. 2023 Oct;597(20):2519-2533. doi: 10.1002/1873-3468.14749. Epub 2023 Oct 15. PMID 37795679
- [Background] Stewart M. Polyadenylation and nuclear export of mRNAs. J Biol Chem. 2019 Mar 1;294(9):2977-2987. doi: 10.1074/jbc.REV118.005594. Epub 2019 Jan 25. PMID 30683695